CLINICAL TRIAL: NCT06925165
Title: Ultrasound Measured Hyomental Distance to Tongue Thickness Ratio as a Predictor of Difficult Intubation in Infants
Status: Active, not recruiting | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Other Study IDs: FMASU MS 53/2025
Record Dates: First submitted 2025-03-06; First posted 2025-04-13 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-03

CONDITIONS: Ultrasound

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Evaluation the role of ultrasound measured hyomental distance to tongue thickness ratio in predicting difficult intubation in infants

DETAILED DESCRIPTION:
Sonographic assessment of the airway after induction of anesthesia and Master Degree Thesis / MFA/ISRO/ Faculty Of Medicine/ASU Page 6 intubation: All infants will be placed in a supine position with their heads slightly extended. Then, the low-frequency probe (curved) will be first placed under the chin in the midsagittal plane and adjusted to show a clear view of the entire tongue outline and the border of the mandible and hyoid bone on the screen. The image will be frozen and stored. On the image the tongue thickness will be measured, which is the maximum vertical distance from the sub mental skin to the tongue surface (Yao W, Wang B 2017). After that, the HMDE will be measured, which is the distance from the lower border of the mentum of the mandible to the upper border of the hyoid bone.

ELIGIBILITY:
Inclusion Criteria:

* Infants aged 1 to 12 months

Both sexes.

Physical status ASA I or II

Exclusion Criteria:

* Restricted mobility of temporomandibular joint
* Absent anesthesia or surgical consent
* Maxillofacial trauma or tumors
* A large mass or scar under the chin

Ages: 1 Month to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Infants aged 1 to 12 months
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2025-01-29 (Actual); Primary Completion 2025-07-29 (Estimated); Study Completion 2025-07-29 (Estimated)

PRIMARY OUTCOMES:
role of ultrasound measured hyomental distance to tongue thickness ratio in predicting difficult intubation in infants. | 2 to 3 minutes after induction of anaesthesia and intubation
  Difficult intubation can be a significant life threatening problem in anesthesia which can lead to serious complications like hypoxia, aspiration, esophageal intubation, emergency surgical airway, cardiovascular instability, cardiac arrhythmias, ischemic encephalopathy, and death.
  In the study investigators will use hyomental distance and tongue thickness measured by ultrasound to suspect difficult intubation in infants aged 1 to 12 month.

CONTACTS AND LOCATIONS:
Overall Officials: Shaimaa Reda Ahmed, MBBCH, Principal Investigator — Anesthesia resident Ain Shams University
Locations (1):
- Ain Shams University, Cairo, Egypt, Egypt

IPD SHARING:
Plan to Share IPD: Yes
all data will be shared once study is completed
Time Frame: before 1/2026
Access Criteria: free